CLINICAL TRIAL: NCT07275567
Title: Data-driven Development of a Core Dataset for Documentation of Difficult Airway Alerts - a Secondary Analysis of Pooled Database From Three Prospective Studies - the FingAIRprint Project
Brief Title: Data-driven Development of a Core Dataset for Difficult Airway Alerts
Acronym: FingAIRprint
Status: Active, not recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-300503-WF
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Airway Management; Intubation; Difficult or Failed; Airway Complication of Anesthesia
Keywords: Difficult airway alerts; Airway alert cards; Airway documentation; Electronic health records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous difficult airway management is the most accurate predictor of future difficulty. Consistent documentation is paramount for future airway planning, but requires reliable, reproducible and easily accessible information. Currently, anaesthesia alert cards are often based on analogue hard copies while they lack a clinically meaningful core data set allowing structured reproducible documentation and risk estimation. Further, existing alert cards are often inconsistently used and clear triggers for issuing of airway alert cards are widely undefined. The FingAIRprint project aims to develop a justifiable core data set using a data-driven approach in patients undergoing tracheal intubation with videolaryngoscopy or direct laryngoscopy, that is intended to be used for documentation of digital airway alerts.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia with tracheal intubation
* Informed consent obtained
* Age > 18 years

Exclusion Criteria:

* Indication for intubation via a bronchoscope or awake intubation
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pooled database from three prospective studies originating from a single study center in adults undergoing elective head and neck surgery with general anaesthesia and tracheal intubation.
Sampling Method: Probability Sample
Enrollment: 1785 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Difficult airway alert | 1 hour
  Documented by the airway operator following tracheal intubation (y/n)

SECONDARY OUTCOMES:
Recommendation for awake tracheal intubation | 1 hour
  Recommendation for future airway planning documented by the airway operator after tracheal intubation (y/n)
Recommendation for camera-assisted tracheal intubation | 1 hour
  Recommendation for future airway planning documented by the airway operator after tracheal intubation (y/n)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Center for Anesthesiology and Intensive Care Medicine, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Result] Kohse EK, Siebert HK, Sasu PB, Loock K, Dohrmann T, Breitfeld P, Barclay-Steuart A, Stark M, Sehner S, Zollner C, Petzoldt M. A model to predict difficult airway alerts after videolaryngoscopy in adults with anticipated difficult airways - the VIDIAC score. Anaesthesia. 2022 Oct;77(10):1089-1096. doi: 10.1111/anae.15841. Epub 2022 Aug 25. PMID 36006056
- [Result] Kohl V, Wunsch VA, Muller MC, Sasu PB, Dohrmann T, Peters T, Tolkmitt J, Dankert A, Krause L, Zollner C, Petzoldt M. Hyperangulated vs. Macintosh videolaryngoscopy in adults with anticipated difficult airway management: a randomised controlled trial. Anaesthesia. 2024 Sep;79(9):957-966. doi: 10.1111/anae.16326. Epub 2024 May 24. PMID 38789407
- [Result] Popal Z, Sieg HH, Muller-Wiegand L, Breitfeld P, Dankert A, Sasu PB, Wunsch VA, Krause L, Zollner C, Petzoldt M. Decision-Making Tool for Planning Camera-Assisted and Awake Intubation in Head and Neck Surgery. JAMA Otolaryngol Head Neck Surg. 2025 Jun 1;151(6):585-594. doi: 10.1001/jamaoto.2025.0538. PMID 40310618